CLINICAL TRIAL: NCT04014153
Title: The Impact of Comorbidity as a Risk Factor of Acute Kidney Injury (AKI) in Patients With Stable Coronary Artery Disease (CAD)
Brief Title: CI-AKI in Patients With Stable CAD and Comorbidities. Are we Doing Better?
Status: Completed | Type: Observational
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Principal Investigator, Olga Mironova, Principal Investigator, I.M. Sechenov First Moscow State Medical University
Other Study IDs: 1/13
Record Dates: First submitted 2019-07-07; First posted 2019-07-10 (Actual); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: Stable Angina; Acute Kidney Injury; Contrast-induced Nephropathy
Keywords: acute kidney injury; coronary artery disease; contrast-induced acute kidney injury; comorbidity; CI-AKI; stable CAD
MeSH Terms: conditions — Angina, Stable; Acute Kidney Injury; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1 (5-year prognosis)
  Interventions: Procedure: Iodinated contrast media
- Group 2 (1-year prognosis)
  Interventions: Procedure: Iodinated contrast media

INTERVENTIONS:
Procedure: Iodinated contrast media — Percutaneous coronary intervention with iodinated contest media

SUMMARY:
Patients aged 18-89 with stable CAD and comorbidities receiving optimal medical treatment requiring PCI with iodinated contrast media.

The aim of the study is to assess the prevalence of contrast-induced AKI in 2012-2013 and 2017 cohorts and to evaluate the potential risk factors of CI-AKI to better guide the prevention in patients of higher risk.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Male and female patients 18 y. o. and older
* Verified stable coronary artery disease (CAD)
* Receiving optimal medical treatment and requiring percutaneous coronary intervention (PCI) with iodinated contrast media

Exclusion Criteria:

* Pregnancy, lactation
* Conditions affecting the prognosis (kidney failure, liver failure, oncology)
* Acute coronary syndrome (ACS)
* Stroke
* Contraindications to PCI
* Therapy with nephrotoxic drugs during the enrolment which cannot be stopped
* Refusal to sign the informed consent

Ages: 18 Years to 89 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Both genders suffering from stable coronary artery disease, requiring percutaneous coronary intervention with intra-arterial iodinated contrast injection
Sampling Method: Probability Sample
Enrollment: 1023 (Actual)
Dates: Start 2012-05-16 (Actual); Primary Completion 2017-10-19 (Actual); Study Completion 2018-12-12 (Actual)

PRIMARY OUTCOMES:
Overall mortality | 5 years
Cardiovascular mortality | 5 years
Myocardial infarction | 5 years
Stroke | 5 years
GI bleeding | 5 years
CABG | 5 years
  CABG after PCI at enrolment
PCI | 5 years
  Repeat PCI after the enrolment

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mironova OIu. [Contrast substances-induced nephropathy]. Ter Arkh. 2013;85(6):90-5. Russian. PMID 23875199
- [Derived] Mironova OI, Deev AD, Lakotka PG, Fomin VV. [Anemia as a risk factor of contrast-associated acute kidney injury]. Ter Arkh. 2020 Dec 15;92(12):48-52. doi: 10.26442/00403660.2020.12.200450. Russian. PMID 33720573
- [Derived] Mironova OI, Staroverov II, Sivakova OA, Deev AD, Fomin VV. [Contrast-induced acute kidney injury in chronic coronary artery disease patients with diabetes mellitus and obesity]. Ter Arkh. 2020 Nov 24;92(10):29-33. doi: 10.26442/00403660.2020.10.000753. Russian. PMID 33346476